CLINICAL TRIAL: NCT01612715
Title: Analysis of Fel d 1-specific T Cells After Airway Allergen Challenge in Asthma:Frequency and Phenotype and Trafficking of Cat Allergen-specific T-cells in Blood, Bone Marrow and Bronchoalveolar Lavage Fluid (BALF) Following Segmental Allergen Challenge in Allergic Asthma.
Brief Title: Analysis of Fel d 1-specific T Cells After Airway Allergen Challenge in Asthma
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Gail Gauvreau, Associate Professor, Hamilton Health Sciences Corporation
Other Study IDs: HHS-12-197
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Allergic Asthma
Keywords: Asthma, allergen challenge, T cells, Fel d 1.
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Population: Mild asthma, cat-allergic, 18-65 years old, males and females will be recruited for the study.
  Interventions: Other: Segmental Allergen Challenge

INTERVENTIONS:
Other: Segmental Allergen Challenge — segmental allergen challenge

SUMMARY:
Cat allergies are a major trigger of asthma. Therapies are being developed to control the allergic response to cats. We are interested in measuring a type of white blood cell which is linked to cat allergies, which will help us understand how to use new therapies in people who suffer from cat allergies and asthma. We will study cat-allergic individuals with stable, mild asthma who will be exposed to cat allergens. We will measure various white blood cells, including the cells that are linked to cat allergies, to determine whether the number of these cells changes following cat exposure. These cells will be measured from the blood and bone marrow by removing samples using a needle. These cells will also be measured from the lungs by inserting a bronchoscope into the airways and drawing up fluid containing cells. This study will improve our understanding of the harmful versus protective role of these cat-specific cells, and will allow for development of better drugs for treatment of asthma triggered by cat exposure.

ELIGIBILITY:
INCLUSION CRITERIA:

1) Male or female, aged 18-65 years. (2) Asthmatic subjects with mild allergic asthma. (3) Positive skin prick test to cat allergen with a wheal diameter at least 2mm l. (4) RAST score of at least 1 or equivalent international units/mL.

(5) Subjects must express one (or more) of the following Human Leukocyte Antigens (HLA): HLA-DRB1*0101, HLA-DRB1*0301, HLA-DRB1*0401, HLA-DRB1*0405, HLA-DRB1*0701, HLA-DRB1*0901, HLA-DRB1*1001, HLA-DRB1*1101, HLA-DRB1*1301, HLA-DRB1*1401, HLA-DRB5*0101.

(6) Methacholine provocative concentration causing a 20% fall in the FEV1 (PC20) > 0.125 mg/ml and <16 mg/mL.

(7) Development of early asthmatic response (≥20% fall in FEV1) with or without a late phase asthmatic response during a screening whole lung allergen challenge.

(8)Willing and able to provide written informed consent. (9) The subject must be willing and able to comply with the study requirements. (10) If the subject is female and of childbearing potential she must practice an acceptable form of contraception, and produce a negative urine pregnancy test on the Screening Visit and at Days -27 and 1. A female subject may be included without a negative urine pregnancy test if she can document that she is surgically sterile or at least 2 years post-menopausal.

(11) Normal chest Xray within 1 year of the screening period

EXCLUSION CRITERIA

1) A history of anaphylaxis to cat allergen. (2) Subjects with an FEV1 <70% of predicted and an FEV1/FVC ratio of < 70. (3) Receipt of any allergen immunotherapy within the last 10 years.

(4) Use of inhaled or nasal corticosteroids or regular antihistamine use or any regular medication to manage asthma.

(5) Subjects for whom administration of epinephrine is contra-indicated (e.g. subjects with acute or chronic symptomatic coronary heart disease or severe hypertension).

(6) Subjects being treated with beta-blockers. (7) Symptoms of a clinically relevant illness, in the Investigator's opinion, within 6 weeks prior to Screening Visit.

(8) Female subjects who are pregnant, lactating or planning a pregnancy during the study.

(9) Any clinically relevant abnormalities detected on physical examination. (10) Vital signs (blood pressure, pulse rate, respiratory rate, body temperature) that are outside normal limits, unless the abnormality is considered not to be of clinical relevance by the Investigator.

(11) Laboratory values (haematology, biochemistry, urine tests) that are outside the normal ranges, unless the abnormality is considered not to be of clinical relevance by the Investigator.

(12) History of alcohol or drug abuse that in the opinion of the Principal Investigator could significantly affect the outcomes of this study.

(13) History of any immunopathological diseases which may confound study outcomes.

(14) History of vasovagal reaction in the last 10 years associated with venipuncture.

(15) Received treatment with an investigational drug within 3 months prior to study.

(16) Unable to communicate or to understand the requirements of the study, which would impair communication between the subject and the Investigator thereby interfering with the informed consent procedure or the gathering of study data.

(17) A history of any significant disease or disorder (e.g. autoimmune, cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, neoplastic/malignant, psychiatric, major physical impairment, severe atopic dermatitis) which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results of the study, or the subject's ability to participate in the study.

(18) Positive test results for Hepatitis B, Hepatitis C, HIV other than would be anticipated following vaccination or history of tuberculosis.

(19) Asthma exacerbation or lower respiratory tract infection in the past 6 weeks.

(20) Subject who has donated blood (including blood products) or experienced loss of blood ≥ 500 mL within 2 months of study screening (21) Subject who has regularly used nicotine or tobacco containing products (including but not limited to: snuff, chewing tobacco, cigars, cigarettes, pipes, or nicotine patches) during 12 months before enrollment/randomization and during the study. A subject who is a former smoker and has smoked >10 pack years must be excluded.

(22) Subject is unwilling to avoid rigorous exercise and caffeinated beverages for at least 4 hours before study visits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mild asthma, cat-allergic, 18-65 years old, males and females will be recruited for the study.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2014-01-29 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
Comparison | 5 Years
  The primary outcome for Aim 1 of the study is to compare the number of tetramer+ T cells in the airways of early and dual-responder subjects after segmental allergen challenge. The primary outcome for Aim 2 of the study is to compare the number of tetramer+ T cells in the bone marrow of early and dual-responder subjects after segmental allergen challenge. This will be measured using a panel of antibodies and flow cytometric analysis of cell surface markers.

SECONDARY OUTCOMES:
Measurements | 5 Years
  The secondary outcome is to determine the frequency, memory phenotype and chemokine receptor profile of tetramer+ T cells in the peripheral blood before and after bronchial allergen challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Gail Gauvreau, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada